CLINICAL TRIAL: NCT07350564
Title: Intensive Blood Pressure Control After Endovascular Thrombectomy for Acute Embolic Stroke (INTENSE): a Multicentre, Open-label, Blinded-endpoint, Randomised Controlled Trial
Brief Title: Intensive Versus Conventional Blood Pressure Control Following Stroke Thrombectomy
Acronym: INTENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hao Yonggang (Other)
Responsible Party: Sponsor-Investigator, Hao Yonggang, Vice Chair of Neurology, The Fourth Affiliated Hospital of Soochow University
Organization: The Fourth Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240024
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: stroke; endovascular thrombectomy; blood pressure; randomised controlled trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive blood pressure target group (Experimental)
  Interventions: Other: Intensive blood pressure management
- Standard blood pressure target group (Active Comparator)
  Interventions: Other: Conventional blood pressure management

INTERVENTIONS:
Other: Intensive blood pressure management — The objective is to achieve a systolic blood pressure (SBP) <120 mmHg within 1 hour after randomization and maintain this target for 48 hours. Intravenous titration is initiated immediately after randomization, with an SBP of 100 mmHg used as the threshold for discontinuing antihypertensive therapy or initiating vasopressors.
  Arms: Intensive blood pressure target group
Other: Conventional blood pressure management — The objective is to maintain an SBP of 140-180 mmHg within 1 hour after randomization and sustain this range for 48 hours. Intravenous antihypertensive agents are administered when SBP exceeds 180 mmHg and discontinued once SBP is ≤150 mmHg.
  Arms: Standard blood pressure target group

SUMMARY:
This clinical trial aims to investigate the safety and efficacy of intensive blood pressure lowering after successful reperfusion with thrombectomy in patients with acute anterior circulation large artery occlusive stroke. The main questions it aims to answer are:

What is the optimal blood pressure range after revascularization with thrombectomy in patients with cerebral embolism? Can intensive blood pressure lowering improve outcomes in cerebral embolism patients following thrombectomy?

Participants will be randomly assigned to either the intervention group, which receives stricter blood pressure control (systolic blood pressure target <120 mmHg), or the control group, which follows a conventional blood pressure management approach (systolic blood pressure target 140-180 mmHg). Outcomes will be assessed during a 3-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* To receive endovascular thrombectomy <24 hours after the onset of symptoms
* Diagnosed with acute anterior circulation ischemic stroke
* National Institutes of Health Stroke Scale (NIHSS) score ≤ 30;
* Alberta Stroke Program Early CT Score (ASPECTS) ≥ 6
* Computed Tomography Angiography (CTA), Magnetic Resonance Angiography (MRA), or Digital Subtraction Angiography (DSA) confirming occlusion of the intracranial internal carotid artery or M1/M2 segment of the middle cerebral artery
* Successful recanalization of the occluded vessel without in-situ or proximal stenosis (modified Treatment in Cerebral Infarction, mTICI ≥ 2b)
* Sustained elevated systolic blood pressure (≥140 mmHg for at least two consecutive measurements, separated by >10 minutes) within 3 hours of reperfusion
* Written informed consent provided by the patient or their legal representative

Exclusion Criteria:

* Pre-existing stroke disability defined by a modified Rankin score (mRS) >2
* Unlikely to benefit from or tolerate endovascular thrombectomy, such as severe allergic reaction to contrast agents
* Failure to achieve mTICI ≥ 2b with endovascular intervention, or presence of in situ or proximal vascular stenosis
* Patients with contraindications for the use of antihypertensive medications, such as allergy to components
* Intracranial space-occupying lesions, including brain tumors and vascular malformations
* Patients with severe liver or renal dysfunction, or those receiving dialysis (severe liver dysfunction is defined as alanine aminotransferase [ALT] > 3 times the upper limit of normal or aspartate aminotransferase [AST] > 3 times the upper limit of normal; severe renal dysfunction is defined as serum creatinine > 3.0 mg/dL [265.2 μmol/L] or glomerular filtration rate [GFR] < 30 mL/min/1.73 m²)
* Serious illness with life expectancy of <6 months
* Lactating women
* Participation in other interventional clinical trials within the past 3 months;
* Any other conditions that render patients unsuitable for participation in this study or unable to complete the study process, such as psychiatric disorders, cognitive or emotional impairments, or physical conditions that hinder compliance with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence at 3 months | At 90 days after randomization
  A modified Rankin Scale (mRS) score of 0 to 2
Symptomatic intracerebral hemorrhage | At 24±12 hours after randomization
  Defined by the Heidelberg Bleeding Classification criteria
All-cause mortality | At 90 days after randomization

SECONDARY OUTCOMES:
Excellent outcome | At 90 days after randomization
  A modified Rankin Scale (mRS) score of 0 to 1
Serious adverse outcome | At 90 days after randomization
  A modified Rankin Scale (mRS) score of 5 to 6
Shift in scores on the mRS | At 90 days after randomization
Infarct volume at follow-up CT scan (24±12h) | At 24±12 hours after randomization
NIHSS score at 24 hours | At 24 hours after randomization
Change in National Institute of Health Stroke Scale (NIHSS) at 24 hours | At 24 hours after randomization
Excellent recovery of NIHSS score at 24 hours | At 24 hours after randomization
  NIHSS 0-1 or improvement of more than 8
Change in National Institute of Health Stroke Scale (NIHSS) at 7 days | At 7 days after randomization
Edema volume assessed by CT | At 7 days after randomization
Health-related quality of life (EQ-5D-3L index score) | At 90 days after randomization
  Health-related quality of life assessed using the EuroQol EQ-5D-3L descriptive system, converted to an index score using [country]-specific value set.
Health-related quality of life (EQ-5D VAS) | At 90 days after randomization
  Self-rated health status assessed using the EuroQol visual analog scale (EQ-VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Asymptomatic ICH | At 24±12 hours after randomization
Large cerebral infarction or intracranial hemorrhage requiring neurosurgical intervention | At 7 days after randomization
Extracranial hemorrhage | An 7 days after randomization
  Examples include gastrointestinal bleeding, urinary tract bleeding, oral or nasal mucosal bleeding, and subcutaneous hematoma.
Non-hemorrhagic serious adverse events | At 7 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

DOCUMENTS (1):
  • Study Protocol (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT07350564/Prot_000.pdf